CLINICAL TRIAL: NCT02962102
Title: Activated Vitamin D for the Prevention and Treatment of Acute Kidney Injury (ACTIVATE-AKI)
Brief Title: Activated Vitamin D for the Prevention and Treatment of Acute Kidney Injury
Acronym: ACTIVATE-AKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Leaf (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David Leaf, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016P002527; 5K23DK106448 (NIH)
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Critically Ill; Acute Kidney Injury
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury | interventions — Calcifediol; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Calcifediol (Experimental): Calcifediol 400mcg orally x 1, followed by 200mcg orally daily x 4
  Interventions: Drug: Calcifediol
- Calcitriol (Experimental): Calcitriol 4mcg orally daily x 5 days
  Interventions: Drug: Calcitriol
- Placebo (Placebo Comparator): Equal volume of medium chain triglyceride (MCT) oil orally daily x 5 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Calcifediol — Calcifediol 400mcg orally x 1, followed by 200mcg orally daily x 4
  Arms: Calcifediol
Drug: Calcitriol — Calcitriol 4mcg orally daily x 5
  Arms: Calcitriol
Drug: Placebos — Placebo (medium chain triglyceride oil) orally daily x 5
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of calcifediol (25-hydroxyvitamin D) and calcitriol (1,25-dihydroxyvitamin D) in preventing and reducing the severity of acute kidney injury (AKI) in critically ill patients.

DETAILED DESCRIPTION:
Decreased circulating levels of active vitamin D metabolites, including 25-hydroxyvitamin D (25D) and 1,25-dihydroxyvitamin D (1,25D), are common in critically ill patients, and lower levels are independently associated with a higher risk of acute kidney injury (AKI). Further, administration of 25D and 1,25D attenuates AKI in animal models. The purpose of this study is to assess if administration of 25D and 1,25D decreases the incidence and severity of AKI in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Admitted to the ICU within 48h prior to enrollment
* Likely to remain in the ICU (alive) for ≥72h
* Naso/orogastric tube or ability to swallow
* High risk of severe AKI

Exclusion Criteria:

* Serum total calcium > 9.0 mg/dl or phosphate > 6.0 mg/dL within previous 48h
* Currently receiving oral calcium supplementation
* Ingestion of vitamin D3 >1,000 IU/day or any 25-hydroxyvitamin D or 1,25-dihydroxyvitamin D during the previous 7 days
* AKI stage 2 or 3 (based on KDIGO serum creatinine and/or urine output criteria)
* History of transplantation or receiving chronic (>7days) of immunosuppressive medications (not including glucocorticoid steroids at a dose less than or equivalent to prednisone 20 mg/day)
* Neutropenia in the previous 48h
* Active primary parathyroid disease, active granulomatous disease, or symptomatic nephrolithiasis in the previous 3 months
* Receiving cytochrome P450 inhibitors
* Chronic Kidney Disease stage V or End Stage Renal Disease
* Hemoglobin < 7 g/dL
* GI malabsorption
* Prisoner
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Leaf, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leaf DE, Shenoy T, Zinchuk K, Gupta S, Dias JA, Sanchez-Almanzar D, Ginde AA, Athar H, Cheng C, Tamura T, Kim EY, Waikar SS. Randomized trial of activated vitamin D for acute kidney injury prevention in critically ill patients. JCI Insight. 2025 Sep 9;10(20):e193523. doi: 10.1172/jci.insight.193523. eCollection 2025 Oct 22. PMID 40924491

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcifediol | Calcitriol | Placebo
Started | 51 | 50 | 49
Completed | 51 | 50 | 49
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcifediol | Calcitriol | Placebo | Total
Number analyzed (Participants) | 51 | 50 | 49 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [53 to 72] | 65 [53 to 74] | 65 [51 to 71] | 65 [52 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 18 | 58
  Male | 32 | 29 | 31 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 11
  Not Hispanic or Latino | 45 | 45 | 46 | 136
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 3 | 15
  White | 43 | 40 | 41 | 124
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 1 | 3
Baseline estimated glomerular filtration rate (eGFR) [Median (Inter-Quartile Range); unit: ml/min/1.73m^2] — Calculated based on the Chronic Kidney Disease-Epidemiology Collaboration equation
  ml/min/1.73m^2 | 94 [77 to 118] | 98 [72 to 121] | 94 [78 to 109] | 95 [75 to 117]
APACHE II score [Median (Inter-Quartile Range); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II (APACHE II), an intensive care unit severity of illness scoring system ranging from 0 to 71, with higher scores indicating more severe disease
  units on a scale | 26 [21 to 30] | 25 [21 to 31] | 27 [22 to 30] | 25 [21 to 30]
Invasive mechanical ventilation [Count of Participants; unit: Participants] | 41 | 43 | 41 | 125
Vasopressors/inotropes [Count of Participants; unit: Participants] | 28 | 28 | 30 | 86
Acute kidney injury [Count of Participants; unit: Participants] — Defined as an increase in serum creatinine ≥0.3 mg/d within the previous 48 hours, ≥50% within the previous 7 days, or urine output ≤0.5 ml/kg/h for 6 consecutive hours
  Participants | 19 | 18 | 18 | 55
Plasma 25-hydroxyvitamin D [Median (Inter-Quartile Range); unit: ng/ml] | 18.8 [11.2 to 26.0] | 17.3 [10.5 to 28.4] | 14.5 [9.7 to 23.0] | 16.5 [10.2 to 26.0]

OUTCOME MEASURES:

1. Primary Outcome: Death Within 7 Days
Description: All-cause mortality within 7 days following randomization
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Calcifediol: Calcifediol 400mcg PO/NGT/OGT x 1, followed by 200mcg PO/NGT/OGT daily x 4
  Calcifediol: Calcifediol 400mcg PO/NGT/OGT x 1, followed by 200mcg PO/NGT/OGT daily x 4
- Calcitriol: Calcitriol 4mcg PO/NGT/OGT daily x 5 days
  Calcitriol: Calcitriol 4mcg PO/NGT/OGT daily x 5
- Placebo: Equal volume of medium chain triglyceride (MCT) oil daily x 5 days
  Placebos: Placebo (medium chain triglyceride oil) daily x 5
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
Participants | 4 | 9 | 6
Statistical Analysis 1: Comparison: Calcifediol vs Placebo; Test type: Superiority; p = 0.52, Fisher Exact
Statistical Analysis 2: Comparison: Calcitriol vs Placebo; Test type: Superiority; p = 0.58, Fisher Exact

2. Primary Outcome: Number of Participants Who Received Renal Replacement Therapy Within 7 Days
Description: Number of participants who received renal replacement therapy within 7 days following randomization
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
Participants | 1 | 1 | 4
Statistical Analysis 1: Comparison: Calcifediol vs Placebo; Test type: Superiority; p = 0.20, Fisher Exact
Statistical Analysis 2: Comparison: Calcitriol vs Placebo; Test type: Superiority; p = 0.20, Fisher Exact

3. Primary Outcome: Relative Average Change in Serum Creatinine From Day 0 to Days 1-7
Description: Average percentage change in serum creatinine assessed on days 1-7 as compared to day 0
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: Relative average percent increase
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
Relative average percent increase | -2.3 [-20.7 to 18.3] | -7.1 [-18.1 to 12.3] | -7.4 [-21.5 to 10.4]
Statistical Analysis 1: Comparison: Calcifediol vs Placebo; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Calcitriol vs Placebo; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With New or Worsening Stage of AKI, Defined by KDIGO Guidelines
Description: Any of the following: 1) an increase in serum creatinine ≥50% compared to the immediate pre-randomization value; 2) new or progressive stage of oliguria; or 3) receipt of renal replacement therapy. Oliguria stages 1, 2, and 3 are defined as urine output (UOP) <0.5 ml/kg/h for 6-12h, <0.5 ml/kg/h for >12h, and <0.3 ml/kg/h for ≥24h or anuria for ≥12h, respectively.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
Participants | 20 | 23 | 19

5. Secondary Outcome: Peak Serum Creatinine (mg/dl)
Description: Highest serum creatinine value on days 1 to 7
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
mg/dl | 1.2 [0.8 to 1.5] | 1.3 [0.8 to 1.9] | 1.2 [0.9 to 1.8]

6. Secondary Outcome: 28-day Mortality
Description: All-cause mortality assessed during the 28 days following randomization
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
Participants | 10 | 16 | 10

7. Secondary Outcome: ICU- and Hospital-free Days
Description: 28 minus the number of days in the ICU or hospital, with 0 assigned to patients who die before 28 days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Calcifediol | Calcitriol | Placebo
Number analyzed (Participants) | 51 | 50 | 49
Days
  ICU-free days | 20 [2 to 25] | 16 [0 to 25] | 11 [0 to 22]
  Hospital-free days | 5 [0 to 17] | 4 [0 to 15] | 0 [0 to 15]

8. Other Pre Specified Outcome: Kidney Injury - Subgroup Analysis Based on Time Zero 25-hydroxyvitamin D Level Above Versus Below the Median
Description: Composite of daily serum creatinine, need for renal replacement therapy (RRT), or death within 7 days
Time Frame: 7 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Kidney Injury - Subgroup Analysis Based on the Presence or Absence of AKI on Enrollment
Description: Composite of daily serum creatinine, need for renal replacement therapy (RRT), or death within 7 days
Time Frame: 7 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Kidney Injury - Subgroup Analysis Based on APACHE II Score on Enrollment Above Versus Below the Median
Description: Composite of daily serum creatinine, need for renal replacement therapy (RRT), or death within 7 days
Time Frame: 7 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Kidney Injury - Subgroup Analysis Based on ICU Type (Medical Versus Surgical)
Description: Composite of daily serum creatinine, need for renal replacement therapy (RRT), or death within 7 days
Time Frame: 7 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Kidney Injury - Subgroup Analysis Based on the Presence or Absence of Sepsis on Enrollment
Description: Composite of daily serum creatinine, need for renal replacement therapy (RRT), or death within 7 days
Time Frame: 7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days for hypercalcemia and 28 days for all-cause mortality
Arm/Group | Calcifediol | Calcitriol | Placebo
All-Cause Mortality (participants affected / at risk) | 10/51 | 16/50 | 10/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 1/51 | 1/50 | 0/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcifediol (N=51) | Calcitriol (N=50) | Placebo (N=49)
Hypercalcemia (Endocrine disorders) | 1 | 1 | 0 — Serum calcium >10.7 mg/dl within 7 days following randomization

LIMITATIONS AND CAVEATS:
Limited sample size and AKI event rate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT02962102/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT02962102/ICF_001.pdf